CLINICAL TRIAL: NCT04000412
Title: A Novel Myocardial Impedance Mapping System for Ablation of Post-infarction Ventricular Arrhytmias in Humans
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Universitat Politècnica de Catalunya (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-IMS-2015-90
Record Dates: First submitted 2019-06-17; First posted 2019-06-27 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Ventricular Arrythmia; Infarction, Myocardial
Keywords: electrical impedance; cardiac radiofrequency ablation
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CASE GROUP: patients with chronic infarction undergoing catheter ablation of ventricular arrhythmias
  Interventions: Device: CardioZ multifrequency impedance recording system

INTERVENTIONS:
Device: CardioZ multifrequency impedance recording system — Patients will be submitted to mapping of both voltage and tissue impedance. The accuracy of the two maps identifying the extent and transmurality of the infarction will be assesssed by gadolinium imaging.
  Other Names: Cardio-Z

SUMMARY:
Precise identification of the infarct scar is essential for successful catheter ablation of ventricular arrhythmias in patients with chronic myocardial infarction. Voltage mapping of endocardial electrograms is currently used to delineate the necrotic scar but this is influenced by the direction of the activation wave front and is not sensitive enough to differentiate distinct degrees of transmural injury in the scar. Mapping of local myocardial electrical impedance may overcome these limitations.

DETAILED DESCRIPTION:
Clinical series: Patients with chronic infarction undergoing catheter ablation of ventricular arrhythmias will be submitted to mapping of both voltage and tissue impedance. Likewise, the accuracy of the two maps identifying the extent and transmurality of the infarction will be assesssed by gadolinium imaging. The impedance system is already constructed and certified for clinical research use.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 yearts
* Chronic myocardial infarction
* Undergoing ventricular ablation of ventricular arrhythmias

Exclusion Criteria:

* patients with device not suitable for cardiac magnetic ressonance (CMR)
* pregnacy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with chronic myocardial infarction undergoing ablation of ventricular arrhythmias.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2019-03-19 (Actual); Primary Completion 2022-02-04 (Estimated); Study Completion 2022-02-25 (Estimated)

PRIMARY OUTCOMES:
Comparative detection of infarct scar by voltage mapping | 3 hours
  Voltage will be measured at different sites of the infarct scar and healthy tissue.
Comparative detection of infarct scar by impedance mapping | 3 hours
  myocardial local impedance will be measured at different sites of the infarct scar and healthy tissue.
Comparative detection of infarct scar by gadolinium enhanced MR imaging | 30 minutes
  Intensity of gadolinium will be measured at different sites of the infarct scar and healthy tissue.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Amoros-Figueras G, Jorge E, Alonso-Martin C, Traver D, Ballesta M, Bragos R, Rosell-Ferrer J, Cinca J. Endocardial infarct scar recognition by myocardial electrical impedance is not influenced by changes in cardiac activation sequence. Heart Rhythm. 2018 Apr;15(4):589-596. doi: 10.1016/j.hrthm.2017.11.031. Epub 2017 Dec 27. PMID 29197656
- [Background] Jorge E, Amoros-Figueras G, Garcia-Sanchez T, Bragos R, Rosell-Ferrer J, Cinca J. Early detection of acute transmural myocardial ischemia by the phasic systolic-diastolic changes of local tissue electrical impedance. Am J Physiol Heart Circ Physiol. 2016 Feb 1;310(3):H436-43. doi: 10.1152/ajpheart.00754.2015. Epub 2015 Nov 25. PMID 26608340
- [Background] Amoros-Figueras G, Jorge E, Garcia-Sanchez T, Bragos R, Rosell-Ferrer J, Cinca J. Recognition of Fibrotic Infarct Density by the Pattern of Local Systolic-Diastolic Myocardial Electrical Impedance. Front Physiol. 2016 Aug 31;7:389. doi: 10.3389/fphys.2016.00389. eCollection 2016. PMID 27630580